CLINICAL TRIAL: NCT01437085
Title: Quantifying Needle Deflection and Tissue Deformation in Transperineal Interstitial Permanent Prostate Brachytherapy: A Basis for Development of Next-Generation Implant Technique
Brief Title: A Study to Measure Needle Bending and Changes in Prostate Shape During a Prostate Seed Implant
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: 25837
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer
Keywords: Needle deflection; Prostate Deformation; Prostate Brachytherapy; Needles
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prostate brachytherapy is an effective treatment option for men with localized prostate cancer, with excellent cure rates and a favorable toxicity profile. With the current needle insertion technique, seed placement inaccuracy is primarily caused by needle deflection and soft tissue deformation, which both occur during the brachytherapy operation. This study will accrue 20 patients undergoing prostate brachytherapy implants and acquire a series of ultrasound images, video clips and one CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer
* Treated with prostate brachytherapy at the Cross Cancer Institute
* Low and intermediate risk prostate cancer
* ambulatory patients
* stable medical condition
* Over 18 years of age
* Capable of giving informed consent

Exclusion Criteria:

* Any hormonal therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a prostate brachytherapy implant at the Cross Cancer Institute.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-10; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nawaid Usmani, MD, FRCPC, Principal Investigator — University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada